CLINICAL TRIAL: NCT05373290
Title: Adverse Effects and Mechanism of Environmental Endocrine Disrupting Chemicals on Female Reproductive health--the Peking University and Environment Reproductive Health Cohort
Brief Title: A Cohort Study of Environmental Endocrine Disrupting Chemicals and Female Reproductive Health
Acronym: PKU-ERC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Huan, Director of Reproductive Medicine Center, Peking University People's Hospital
Other Study IDs: PKUPHIVF001
Record Dates: First submitted 2022-04-19; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the urine, blood, follicular fluid，semen，villous tissue and placenta
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there is no intervention in the study — there is no intervention in the study

SUMMARY:
Infertility is a disease that seriously affects the physical and mental health of women of childbearing age. The incidence of infertility has been increasing in recent years. Studies have shown that the occurrence of infertility may be related to environmental endocrine disrupting substances. This project was designed to establish a cohort study on environmental endocrine disrupting substances and in vitro fertilization (IVF) treatment, collect blood, urine, semen, follicular fluid, granulosa cells, chorionic decidua biological specimens, and then follow up on the pregnancy outcomes. The concentration of disrupting substances was detected and then found the associations between environmental endocrine disrupting substances and female reproductive health.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of infertile patients undergoing IVF treatment

Exclusion Criteria:

Donor egg transplants excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the couples intended to receive the treatment of IVF can be included in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of eggs retrieved | immediately after the eggs retrieved
  the number of eggs retrieved in the process of in vitro fertilization (IVF)
the number of available embryos | 1 week after the eggs retrieved
  the number of available embryos in the process of IVF
the clinical pregnancy rate | 4 weeks after the embryos transfer
  the clinical pregnancy rate in the process of IVF
the miscarriage rate | 7 months after embryos transfer
  the miscarriage rate in the process of IVF
the live birth rate | 40 weeks after embryos transfer
  the live birth rate in the process of IVF

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Liang Y, Dong X, Fu M, Wang Y, Wang Y, Han H, Wang M, Zuo Y, Zhang S, Shen H, Han F, Gao F. Association between snoring and in vitro fertilization outcomes among infertile women. Sleep Med. 2025 Apr;128:74-81. doi: 10.1016/j.sleep.2025.01.013. Epub 2025 Jan 21. PMID 39892082